CLINICAL TRIAL: NCT04050865
Title: CLN-0052, A Multi-Center, Randomized, Double-Masked, Vehicle Controlled Phase 3 Study Evaluation the Efficacy and Safety of OTX-DP for the Treatment of Allergic Conjunctivitis Using a Modified Conjunctival Allergen Challenge Model (Ora-CAC®)
Brief Title: A Study Evaluating the Safety and Efficacy of OTX-DP for the Treatment of Allergic Conjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLN-Protocol-0052
Record Dates: First submitted 2019-08-07; First posted 2019-08-08 (Actual); Results first posted 2021-10-07 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OTX-DP (Experimental)
  Interventions: Drug: Dexamethasone, 0.4mg
- Placebo (Placebo Comparator)
  Interventions: Device: Placebo plug with no drug

INTERVENTIONS:
Drug: Dexamethasone, 0.4mg — Ophthalmic Insert
  Other Names: OTX-DP
  Arms: OTX-DP
Device: Placebo plug with no drug — Ophthalmic Insert
  Arms: Placebo

SUMMARY:
The objective of the study is to evaluate the efficacy and safety of OTX-DP as a dexamethasone ophthalmic insert when placed in the canaliculus of the eyelid for the treatment of the signs and symptoms of allergic conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* Has a positive history of ocular allergies and a positive skin test reaction to a perennial allergen and a seasonal allergen
* Has a positive bilateral CAC reaction to a perennial allergen within minutes of instillation

Exclusion Criteria:

* History of refractive surgery (including LASIK procedures) within the past 2 years
* History of retinal detachment, diabetic retinopathy, or active retinal disease
* Presence of an active ocular infection or positive history of an ocular herpetic infection at any visit
* History of IOP increase as a result of steroid treatment
* A female who is currently pregnant, planning a pregnancy, or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Vision Institute, Colorado Springs, Colorado
  - The Eye Care Institute, Louisville, Kentucky
  - Andover Eye Associates, Raynham, Massachusetts
  - Silverstein Eye Centers, Kansas City, Missouri
  - Total Eye Care, P.A., Memphis, Tennessee
  - Eye Associates of Texas, Round Rock, Texas

REFERENCES:
- [Derived] Kenyon K, McLaurin EB, Silverstein SM, Meyer JC, Anderson E, Patel RH, Gomes PJ, Reilly E, Vantipalli S, Cheung MW, Goldstein MH. A Randomized, Multicenter Phase 3 Clinical Trial Evaluating Intracanalicular Dexamethasone Insert for the Treatment of Allergic Conjunctivitis. Clin Ophthalmol. 2024 Sep 21;18:2671-2684. doi: 10.2147/OPTH.S476419. eCollection 2024. PMID 39328900

RESULTS

PARTICIPANT FLOW:
Groups:
- OTX-DP, 0.4 mg: OTX-DP, 0.4 mg
- Placebo: Placebo Vehicle
Period: Overall Study
Arm/Group | OTX-DP, 0.4 mg | Placebo
Started | 48 | 48
Completed | 44 | 43
Not Completed | 4 | 5
Not completed — Adverse Event | 1 | 0
Not completed — no insert | 1 | 0
Not completed — Only 1 insert | 2 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- OTX-DP: OTX-DP
- Total: Total of all reporting groups
Arm/Group | OTX-DP | Placebo | Total
Number analyzed (Participants) | 48 | 48 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 45 | 92
  >=65 years | 1 | 3 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (12.45) | 46.0 (12.92) | 44.9 (12.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 24 | 51
  Male | 21 | 24 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 17 | 31
  White | 32 | 29 | 61
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 48 | 48 | 96

OUTCOME MEASURES:

1. Primary Outcome: Ocular Itching Post-CAC (Conjunctival Allergen Challenge) at Visit 6 (7 Days Post-insertion)
Description: Modified CAC model (Ora, Andover, MA); Grade 0-4, allowing half unit Increments; 0 = None 0.5 = An intermittent tickle sensation possibly localized in the corner of the eye 1.0 = An intermittent tickle sensation involving more than just the corner of the eye 1.5 = An intermittent all-over tickling sensation 2.0 = A mild continuous itch (can be localized) without desire to rub 2.5 = A moderate, diffuse continuous itch with desire to rub 3.0 = A severe itch with desire to rub 3.5 = A severe itch improved with minimal rubbing 4.0 = An incapacitating itch with an irresistible urge to rub 0.5 unit increments ARE allowed
Time Frame: 3 minutes
Population: ITT Population with Multiple Imputation (MCMC) Subject Level Imputation
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | OTX-DP | Placebo
Number analyzed (Participants) | 48 | 48
units on a scale | 1.80 [1.51 to 2.08] | 2.69 [2.40 to 2.98]

2. Primary Outcome: Ocular Itching Post-CAC (Conjunctival Allergan Challenge) at Visit 6 (7 Days Post-insertion)
Description: as for outcome 1
Time Frame: 5 minutes
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | OTX-DP | Placebo
Number analyzed (Participants) | 48 | 48
units on a scale | 1.73 [1.45 to 2.00] | 2.72 [2.44 to 3.01]

3. Primary Outcome: Ocular Itching Post-CAC (Conjunctival Allergan Challenge) at Visit 6 (7 Days Post-insertion)
Description: as for outcome 1
Time Frame: 7 minutes
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | OTX-DP | Placebo
Number analyzed (Participants) | 48 | 48
units on a scale | 1.72 [1.43 to 2.00] | 2.71 [2.43 to 2.99]

ADVERSE EVENTS:
Time Frame: 30 Days
Arm/Group | OTX-DP | Placebo
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 16/48 | 14/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OTX-DP (N=48) | Placebo (N=48)
Treatment Emergent Adverse Events (Eye disorders) | 16 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-10-29): https://cdn.clinicaltrials.gov/large-docs/65/NCT04050865/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-27): https://cdn.clinicaltrials.gov/large-docs/65/NCT04050865/SAP_001.pdf